CLINICAL TRIAL: NCT06580184
Title: Theoretically Informed Behavioral Intervention to Prevent HIV-related Comorbidities
Brief Title: Theoretically Informed Behavioral Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000033508; R01MD019956 (NIH)
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: HIV; CVD; Metabolic Disease
Keywords: Syndemic; HIV; CVD; HTN; Diabetes Mellitus; Cancer; Virtual Reality; Prevention
MeSH Terms: conditions — Metabolic Diseases; Diabetes Mellitus; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LEARN 2 Platform (Experimental): The intervention arm in this study involves participants engaging with the LEARN2 virtual environment, designed to provide tailored prevention education for HIV-related comorbidities with shared risk factors. Participants will navigate a virtual platform focused on health education related to body systems, utilizing customizable avatars for anonymity and comfort.
  Interventions: Behavioral: LEARN 2 Platform
- Waitlist Control (Active Comparator): The waitlist control group will not have immediate access to the LEARN2 intervention but will receive a welcome packet with information on how to contact the study team and the date they will gain access to the intervention after a waiting period. This design helps to ensure that all participants eventually receive the intervention while allowing researchers to assess the efficacy of the LEARN2 platform.
  Interventions: Behavioral: LEARN 2 Platform

INTERVENTIONS:
Behavioral: LEARN 2 Platform — The LEARN 2 Platform will provide tailored prevention education of HIV-comorbidities with shared risk factors. Participants will navigate LEARN 2 and access targeted health content.

SUMMARY:
The goal of this waitlist control clinical trial is to learn if the tailored LEARN 2 platform can prevent HIV-related comorbidities with shared risk factors in men ages 18 and older living with HIV. The main question[s] are:

1. Can the virtual environment improve quality of life among these participants?
2. Does the LEARN 2 platform effectively serve as prevention education for HIV comorbidity shared risk factors?

Researchers will compare participants receiving the LEARN2 virtual environment intervention to those in a waitlist control group to see if the intervention leads to improvements in quality of life and reductions in risk factors.

Participants will be asked to:

1. Engage with the virtual environment weekly.
2. Participate in virtual live health educator sessions.
3. Complete daily assessments of personal health behaviors through Ecological Momentary Assessment.

DETAILED DESCRIPTION:
The goal of this waitlist control clinical trial is to determine the efficacy of the tailored LEARN 2 platform in preventing HIV-related comorbidities characterized by shared risk factors. The principal questions this study aims to address are:

1. Can engagement with the virtual environment enhance the quality of life for participants?
2. Is the LEARN 2 platform effective in providing prevention education of shared risk factors associated with HIV comorbidities?

To evaluate these objectives, the investigators will conduct comparisons between participants allocated to the LEARN 2 virtual environment intervention and those assigned to a waitlist control group. This design will facilitate the assessment of whether participation in the LEARN 2 intervention correlates with significant improvements in quality of life metrics (behavioral and psychosocial) and a reduction in associated health risk factors.

Participants will be instructed to:

1. Engage with the virtual environment on a weekly basis, exploring tailored health content designed to address their specific needs.
2. Attend virtual live sessions with health educators, where they will receive real-time education on health issues relevant to their condition and associated lifestyle factors using the American Heart Association's Life's Essential 8 as a behavioral prevention framework.
3. Complete daily assessments of their personal health behaviors using Ecological Momentary Assessment (EMA), capturing real-time data on behavioral trends that may influence their health outcomes.

This systematic approach aims to generate comprehensive data on the impact of the LEARN 2 intervention on both quality of life and the modulation of health-related behaviors among these at-risk populations.

ELIGIBILITY:
Inclusion Criteria:

Self-identify as:

* living with HIV
* English speaking
* Access to a device compatible with LEARN 2

Exclusion Criteria:

- medical history of serious complications such as heart attack, stroke, cognitive impairment, or cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 164 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life scale | Baseline, 3 and 6 months
  29-item scale from the PROMIS® Profile 29 for adults. The quality- of-life questions include physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, and pain intensity over the past 7 days. Each question, except for the pain intensity question, is measured on a 5-point scale.

SECONDARY OUTCOMES:
Diet | Months 1, 3, and 5
  1-item that has participants rate how healthy one's eating was that day and has been validated in EMA studies
Physical Activity | Months 1, 3, and 5
  3 items that assess the number of minutes of light, moderate, and heavy physical activity and has been validated in EMA studies.
Sleep Quality | Months 1, 3, and 5
  1-item that assesses the quality of sleep for the previous night from 1(poor) to 8(extremely rested) and has been validated in EMA
Health Care Utilization | Months 1, 3, and 5
  assesses perceived health needs, whether they have a plan to deal with those needs, and whether they saw a health care provider about those needs
Physical Relationship Health | Months 1, 3, and 5
  4-items that assess whether participants were intimate and type of activity
Smoking | Months 1, 3, and 5
  2-items used in EMA studies that assessed whether the participant smoked and how many cigarettes
Social Support | Months 1, 3, and 5
  3-item scale that assesses the among of emotional, informational, and tangible support received from their social network
Coping | Months 1, 3, and 5
  7-item scale where participants rate whether they used 7 different coping strategies which has been validated in EMA studies.
Social Cohesion | Months 1, 3, and 5
  7-item scale that measures decree of cohesion within a person's neighborhood or community.

CONTACTS AND LOCATIONS:
Overall Officials: S. Raquel Ramos, PhD, MBA, MSN, Principal Investigator — Yale University
Locations (1):
- Yale University, Orange, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramos SR, Reynolds H, Johnson C, Melkus G, Kershaw T, Thayer JF, Vorderstrasse A. Perceptions of HIV-Related Comorbidities and Usability of a Virtual Environment for Cardiovascular Disease Prevention Education in Sexual Minority Men With HIV: Formative Phases of a Pilot Randomized Controlled Trial. J Med Internet Res. 2024 Aug 22;26:e57351. doi: 10.2196/57351. PMID 38924481